CLINICAL TRIAL: NCT07244588
Title: Evaluation of Tumor Bed Cavity Shaving as an Oncologically Safe Alternative to Frozen Section Analysis in Breast-Conserving Surgery
Brief Title: Shaving as an Safe Alternative to Frozen Section Analysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Ezzat Gerges (Other)
Responsible Party: Sponsor-Investigator, Mark Ezzat Gerges, Resident Physician at General surgery department Assiut University Hospital, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBCS as an alternative to FFS
Record Dates: First submitted 2025-11-15; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Early Stage Breast Cancer
Keywords: Breast cancer; Breast conserve surgery; low socioeconomic settings; Shaving; Margin status; Fresh frozen section; Operative time; Safe Alternative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor bed cavity shaving arm (Experimental): Patients undergoing breast-conserving surgery will receive intraoperative tumor bed cavity shaving as an alternative approach to ensure clear surgical margins. Additional cavity shavings will be taken circumferentially after the primary lumpectomy specimen. The outcomes will be compared with standard margin assessment methods.
  Interventions: Procedure: Tumor bed cavity shaving

INTERVENTIONS:
Procedure: Tumor bed cavity shaving — feasible in centers lacking intraoperative pathological facilities.
  * Time saving (significantly reduces the overall operative time).
  * cost-effectiveness.
  * Technically simple (Easy to perform without the need for specialized equipment or advanced facilities).
  * it represents a suitable option in low- to medium-socioeconomic settings, where resources and advanced intraoperative support may be limited.
    * It is expected to demonstrate comparable oncological safety to Intraoperative Frozen Section Analysis (FSA) in achieving margin negativity with Significant reduction anticipated in Positive margin rates&Re-excision frequency&Operative duration and Overall procedural cost.

SUMMARY:
Evaluation of Tumor Bed Cavity Shaving as an Oncologically Safe Alternative to Frozen Section Analysis in Breast-Conserving Surgery and aim of study To assess the oncological safety and practicality of tumor bed cavity shaving also aims to evaluate its impact on operative time and overall cost.

DETAILED DESCRIPTION:
Breast cancer remains the most common malignancy among women worldwide and represents a major health burden. Breast-conserving surgery (BCS) has become the standard of care for early-stage breast cancer, aiming to achieve complete tumor excision with histologically clear margins combined with adjuvant radiotherapy, offers equivalent survival rates to mastectomy in early-stage cases.

. Positive surgical margins are strongly associated with increased rates of local recurrence and frequently necessitate re-excision.

Traditionally, intraoperative frozen section analysis (FSA) has been used to assess margin status. However, this technique has several drawbacks, including:

* Limited availability in many centers.
* Requires high-experienced cytopathologists making it challenging in resource-limited places.
* Adds substantial cost.
* Time consuming (prolonged operative time).

  * Recently, the tumor bed cavity shaving (TBCS) has been introduced as a more practical alternative technique that can reduce the incidence of positive margins without relying on intraoperative pathology.

tumor bed cavity shaving (TBCS) means additional thin layers of tissue approximately 5:10 mm in thickness are removed circumferentially from the cavity walls .

With many advantages:

* feasible in centers lacking intraoperative pathological facilities.
* Time saving (significantly reduces the overall operative time).
* cost-effectiveness.
* Technically simple (Easy to perform without the need for specialized equipment or advanced facilities).
* it represents a suitable option in low- to medium-socioeconomic settings, where resources and advanced intraoperative support may be limited.

  * It is expected to demonstrate comparable oncological safety to Intraoperative Frozen Section Analysis (FSA) in achieving margin negativity with Significant reduction anticipated in Positive margin rates&Re-excision frequency&Operative duration and Overall procedural cost.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years.
* Diagnosed with unifocal, operable invasive breast carcinoma.
* Suitable for breast-conserving surgery. Criteria:

Exclusion criteria:

-Contraindication of Breast-Conserving Surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of positive margins and re-excision within 2 years post-surgery | From time of enrollment of the patient until 2 years post-operative
  Percentage of patients whose surgical pathology shows positive margins, and percentage of patients who undergo re-excision. Assessment will be based on histopathology reports and surgical records.
  Unit of Measure: percentage number of patients Measurement Tool: Histopathological examination (pathology report) for margin status; surgical database/operative logs for re-excision events.

SECONDARY OUTCOMES:
- Cost-effectiveness - Facilities availability - Impact on intraoperative time | From enrollment time of the patient until 2 years post operative
  1. Cost-effectiveness Description: Total direct cost incurred per patient from surgery through 2 years of follow-up, including operative costs, pathology, imaging, and any re-operations.
     Unit of Measure: Currency Measurement Tool: cost-analysis using hospital accounting data.
  2. Facilities availability Description: Frequency of use and availability of required surgical infrastructure during the study period.
     Unit of Measure: Number / proportion (for example, number of surgeries per facility per month, or percentage of scheduled surgeries using the study's protocol) Measurement Tool: Hospital operation records, facility logbooks or administrative databases.
  3. Impact on intraoperative time Description: Difference in surgical duration (minutes) between standard procedure and the procedure under study, if applicable.
  Unit of Measure: Minutes Measurement Tool: Operative records / anesthesia records. Time Frame: from incision to closure.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Thabet, Study Chair — Assiut University
Locations (1):
- Faculty of Medicine Assiut University, Asyut, Egypt